CLINICAL TRIAL: NCT04556006
Title: The Effect of Training Given to Coronary Artery Patients on Disease Management
Brief Title: Disease Management for Coronary Artery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, Uğur Doğan, Lecturer, Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Kilis7AralikU
Record Dates: First submitted 2020-09-03; First posted 2020-09-21 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-03

CONDITIONS: Patient Empowerment; Coronary Artery Disease
Keywords: Training; Disease Management; Nursing; Coronary Artery Disease; Compliance
MeSH Terms: conditions — Patient Participation; Coronary Artery Disease; Patient Compliance | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Single blinded, randomised-control study
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The patients in the control group received only the standard care provided by the clinicians. After the collection of post-test data, the content of the training was also explained to these patients and the study was completed by giving them the training guide.
- Intervention (Active Comparator): The training program was applied by the researcher who also work as an academic nurse. The contact information of the patients was obtained and the contact information of the researcher was also given to the patients. In order to consolidate the information given, the training guide was given to the patients in the intervention group. After the training, the patients in the intervention group were contacted again in the 2nd week by using face-to-face interview and in the 4th-8th and 12th weeks by phone calls. During these interviews, the questions of the patients, if any, were answered and the problems they faced regarding the disease management were tried to be solved. In the last interview, an appointment day was determined to meet face-to-face at home, workplaces or hospital according to the preferences of the patients.
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — The data collection process of the study was carried out in two stages using data collection tools.
  First stage: Personal Information Form and Compliance Questionnaire were applied to all patients in both groups. After anthropometric measurements, Framingham Risk Score was determined. The data collection forms were filled with the patients using face-to-face interview technique. The data collection process lasted for approximately 10-15 minutes. After the data collection, the patients in the intervention group were trained. No training was given to the patients in the control group but they received a "Coronary Artery Disease Management Guide".
  Second stage: 12 weeks after the first interview, the patients were interviewed again face-to-face interview technique and the forms and measurements applied initially were repeated.
  Arms: Intervention

SUMMARY:
This randomized controlled trial was conducted with 58 patients hospitalized in the cardiology clinic of a state hospital. Personal Information Form, Anthropometric measurements, Framingham risk score, and compliance questionnaire (CQ) were used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and over,
* diagnosed with coronary artery disease for at least 2 months,
* no hearing and vision problem,
* no perception and expression deficiency,
* not diagnosed with any psychiatric disease,
* living in Kilis province,
* voluntary to participate in the study.

Exclusion Criteria:

* aged 18 under,
* diagnosed without coronary artery disease for at least 2 months,
* hearing and vision problem,
* perception and expression deficiency,
* diagnosed with any psychiatric disease,
* no living in Kilis province,
* no voluntary to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: uğur doğan, Ph.D, Principal Investigator — Lecturer
Locations (1):
- Kilis 7 Aralık University, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be a plan to make individual participant data available.
Supporting Information: Study Protocol, SAP
Time Frame: 3 months after the study is completed
Access Criteria: All data
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

REFERENCES:
- [Result] Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR Jr, Smith SC Jr, Spertus JA, Williams SV, Anderson JL; American College of Cardiology Foundation/American Heart Association Task Force. 2012 ACCF/AHA/ACP/AATS/PCNA/SCAI/STS guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association task force on practice guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Circulation. 2012 Dec 18;126(25):e354-471. doi: 10.1161/CIR.0b013e318277d6a0. Epub 2012 Nov 19. No abstract available. PMID 23166211
- [Result] Kurcer MA, Ozbay A. [Effects of patient education and counseling about life style on quality of life in patients with coronary artery disease]. Anadolu Kardiyol Derg. 2011 Mar;11(2):107-13. doi: 10.5152/akd.2011.028. Epub 2011 Feb 2. Turkish. PMID 21285019
- [Result] Bitton A, Choudhry NK, Matlin OS, Swanton K, Shrank WH. The impact of medication adherence on coronary artery disease costs and outcomes: a systematic review. Am J Med. 2013 Apr;126(4):357.e7-357.e27. doi: 10.1016/j.amjmed.2012.09.004. PMID 23507208
- [Derived] Dogan U, Ovayolu N. The effect of training on treatment adherence in coronary artery patients: A single-blind randomised controlled trial. J Clin Nurs. 2022 Mar;31(5-6):744-754. doi: 10.1111/jocn.15933. Epub 2021 Jul 6. PMID 34231274

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The training program was applied by the researcher who also work as an academic nurse. The contact information of the patients was obtained and the contact information of the researcher was also given to the patients. In order to consolidate the information given, the training guide was given to the patients in the intervention group. After the training, the patients in the intervention group were contacted again in the 2nd week by using face-to-face interview and in the 4th-8th and 12th weeks by phone calls. In the last interview, an appointment day was determined to meet face-to-face at home, workplaces or hospital according to the preferences of the patients.
  Patient education: The data collection process of the study was carried out in two stages using data collection tools.
  First stage: The forms were applied to all patients in both groups. After anthropometric measurements, framingham risk score was determined. The data collection forms were filled with the patients using face-to-face interview technique. The data collection process lasted for approximately 10-15 minutes. After the data collection, the patients in the intervention group were trained. No training was given to the patients in the control group but they received a "Coronary Artery Disease Management Guide".
  Second stage: 12 weeks after the first interview, the patients were interviewed again face-to-face interview technique and the forms and measurements applied initially were repeated.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 28 | 30
Completed | 28 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: After the data collection, the patients in the intervention group were trained. The training programme is not only more structured training than the standard care programme but also includes patient follow-up at certain periods. Thus, the effect of the given education and follow-up on patient behaviour is monitored. The training programme is consist of information about disease, treatment process, risk factors and coping mechanisms.
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.21 (11.46) | 56.83 (10.74) | 58.46 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Compliance Questionnaire Scores of the Participants
Description: Compliance Questionnaire is a form allowing to investigate 11 different areas such as the use of medication causing maladaptation in disease management in individuals with chronic illnesses, diet, weight loss, limiting physical activity, exercise, coping with stress, alcohol use, smoking, sexual activity problems, caffeine intake and working/job life. In the form allowing Likert-type evaluation, the participant is expected to select one of the options 0 (never), 1 (very rarely), 2 (sometimes), 3 (most of the time) or 4 (always) while expressing his/her compliance level for each adaptation area. The scores corresponding to the given expression are summed and Compliance Questionnaire score for each participant is determined. The score range that can be obtained for each subscale is 0-4. The Compliance Questionnaire total scores is between 0-44. High scores mean a better as it an increase in the compliance level to the disease.
Time Frame: Initially-12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- İntervention: The contact information of the patients was obtained and the contact information of the researcher was also given to the patients. In order to consolidate the information given, the training guide was given to the patients in the intervention group. After the training, the patients in the intervention group were contacted again in the 2nd week by using face-to-face interview and in the 4th-8th and 12th weeks by phone calls. In the last interview, an appointment day was determined to meet face-to-face at home, workplaces or hospital according to the preferences of the patients.
  Patient education: The data collection process of the study was carried out in two stages using data collection tools.
  First stage: Personal Information Form and Compliance Questionnaire were applied to all patients in both groups. After anthropometric measurements, framingham risk score was determined. The data collection forms were filled with the patients using face-to-face interview technique. The data collection process lasted for approximately 10-15 minutes. After the data collection, the patients in the intervention group were trained. No training was given to the patients in the control group but they received a "Coronary Artery Disease Management Guide".
  Second stage: 12 weeks after the first interview, the patients were interviewed again face-to-face interview technique and the forms and measurements applied initially were repeated.
Arm/Group | Control | İntervention
Number analyzed (Participants) | 28 | 30
score on a scale | 22.25 (7.02) | 22.53 (5.48)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Control: The patients in the control group were given only standard care protocol by clinicians
- Intervention: The training programme is not only more structured training than the standard care programme but also includes patient follow-up at cer-tain periods. Thus, the effect of the given education and follow-up on patient behaviour is monitored. The training programme was applied to patients in intervention group by the first author who also works as an academic nurse.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04556006/Prot_SAP_000.pdf